CLINICAL TRIAL: NCT05756790
Title: Couple-Based Motivational Interviewing With Mobile Breathalyzers to Reduce Alcohol Use in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); The City College of New York (Other); Human Sciences Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P0551145; R34AA029649 (NIH)
Record Dates: First submitted 2023-02-21; First posted 2023-03-06 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS; Alcohol Abuse
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Couples will be randomized 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care (No Intervention): Couples in this condition will receive the standard of care for alcohol use in addition to a brief alcohol counseling session modeled after WHO guidelines and Dr. Conroy's intervention in Malawi, which uses participants' baseline AUDIT scores for messaging around alcohol reduction and lasts 5-10 minutes.
- Motivational Interviewing (MI) (Experimental): Couples will have three MI sessions over a 60-day period. These sessions will focus on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
  Interventions: Behavioral: Motivational Interviewing
- Motivational Interviewing Plus Breathalyzer (MI Plus) (Experimental): In addition to three MI sessions, drinkers in this condition will be prompted via SMS message twice per day to use a mobile app and a breathalyzer to test their blood alcohol levels (BAC). Both the drinker and their partner will receive real-time feedback about alcohol use.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Motivational Interviewing plus Breathalyzer

INTERVENTIONS:
Behavioral: Motivational Interviewing — Counseling
  Arms: Motivational Interviewing (MI); Motivational Interviewing Plus Breathalyzer (MI Plus)
Behavioral: Motivational Interviewing plus Breathalyzer — Counseling plus mobile breathalyzer/ app
  Arms: Motivational Interviewing Plus Breathalyzer (MI Plus)

SUMMARY:
This project aims to develop and pilot test an intervention using couple-based motivational interviewing (MI) and mobile breathalyzers to reduce heavy alcohol use with couples living with HIV in South Africa.

DETAILED DESCRIPTION:
This project aims to develop and test an alcohol intervention using couple-based motivational interviewing (MI) and mobile breathalyzers to build dyadic support around drinking in HIV-affected couples in South Africa. Specifically, the study aims to: 1) To develop a couple-based MI intervention with mobile breathalyzer technology to deliver real-time feedback on BAC levels. We will target heavy alcohol users with HIV and enroll their primary partner; 2) to develop and pilot test the study procedures for a future randomized controlled trial (RCT) of the couple-based intervention; and 3) to determine the feasibility and acceptability (F&A) of couple-based MI as a standalone intervention and when combined with mobile breathalyzers to provide real-time feedback and support to couples. We will also conduct qualitative interviews with a subset of 15 couples to contextualize F&A data and refine our procedures. Our goal is to demonstrate a proof-of-concept for the proposed intervention, which if shown to be feasible and acceptable, may provide a scalable intervention to reduce heavy alcohol consumption and improve HIV treatment outcomes for couples in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* in a primary relationship for at least 6 months
* aged 18-49
* have at least one partner (the "index patient") with a positive AUDIT-C screen score
* has been on antiretroviral therapy (ART) for at least 6 months
* has disclosed HIV status to their partner

Exclusion Criteria:

* Report severe intimate partner violence in the past 3 months and/or fear that their safety would be at risk (reported during screening)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Conroy, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Human Sciences Research Council, Pietermaritzburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
There is a plan in place to share data with the NIAAA Data Archive.
Supporting Information: Study Protocol
Time Frame: Data will be uploaded to the NIAAA Data Archive two times per year while data are being collected. It will be available indefinitely.
Access Criteria: Users must apply for and receive permission from the NIH data archive.
URL: https://www.niaaa.nih.gov/research/data-archive-and-resources/niaaa-data-archive

REFERENCES:
- [Background] Conroy AA, McKenna SA, Ruark A. Couple Interdependence Impacts Alcohol Use and Adherence to Antiretroviral Therapy in Malawi. AIDS Behav. 2019 Jan;23(1):201-210. doi: 10.1007/s10461-018-2275-2. PMID 30218319
- [Background] Starks TJ, Millar BM, Doyle KM, Bertone P, Ohadi J, Parsons JT. Motivational interviewing with couples: A theoretical framework for clinical practice illustrated in substance use and HIV prevention intervention with gay male couples. Psychol Sex Orientat Gend Divers. 2018 Dec;5(4):490-502. doi: 10.1037/sgd0000297. Epub 2018 Jun 25. PMID 30581887
- [Background] Woolf-King SE, Conroy AA, Fritz K, Johnson MO, Hosegood V, van Rooyen H, Darbes L, McGrath N. Alcohol use and relationship quality among South African couples. Subst Use Misuse. 2019;54(4):651-660. doi: 10.1080/10826084.2018.1531428. Epub 2018 Nov 8. PMID 30407888
- [Background] Aharonovich E, Stohl M, Cannizzaro D, Hasin D. HealthCall delivered via smartphone to reduce co-occurring drug and alcohol use in HIV-infected adults: A randomized pilot trial. J Subst Abuse Treat. 2017 Dec;83:15-26. doi: 10.1016/j.jsat.2017.09.013. Epub 2017 Sep 29. PMID 29129192
- [Background] Hahn JA, Emenyonu NI, Fatch R, Muyindike WR, Kekiibina A, Carrico AW, Woolf-King S, Shiboski S. Declining and rebounding unhealthy alcohol consumption during the first year of HIV care in rural Uganda, using phosphatidylethanol to augment self-report. Addiction. 2016 Feb;111(2):272-9. doi: 10.1111/add.13173. Epub 2015 Nov 5. PMID 26381193
- [Background] Lauckner C, Taylor E, Patel D, Whitmire A. The feasibility of using smartphones and mobile breathalyzers to monitor alcohol consumption among people living with HIV/AIDS. Addict Sci Clin Pract. 2019 Nov 26;14(1):43. doi: 10.1186/s13722-019-0174-0. PMID 31771655
- [Derived] Msimango L, Butterfield R, Starks TJ, van Heerden A, Neilands TB, Hahn JA, Chibi B, Humphries H, Conroy AA. Couples motivational interviewing with mobile breathalysers to reduce alcohol use in South Africa: a pilot randomised controlled trial of Masibambisane. BMJ Open. 2024 Jan 30;14(1):e083390. doi: 10.1136/bmjopen-2023-083390. PMID 38296300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the community between March 15, 2023 and Nov 11, 2023.
Pre-assignment Details: People living with HIV who screened positive for heavy drinking were recruited with their primary romantic partners, who may or may not have been living with HIV and may or may not have screened positive for heavy drinking.
  93 couples (186 individuals) were consented and randomized. Three couples (6 individuals) were found to be ineligible and thus were excluded from analyses of baseline characterisitcs, outcome measures and adverse events. Ninety couples (180 individuals) were included.
Groups:
- Enhanced Usual Care- Heavy Drinkers: People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. They received the standard of care for alcohol use in addition to a brief alcohol counseling session modeled after WHO guidelines and Dr. Conroy's intervention in Malawi, which uses participants' baseline AUDIT scores for messaging around alcohol reduction and lasts 5-10 minutes. They attended this brief counseling session with their primary romantic partner.
- Enhanced Usual Care (EUC)- Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the EUC arm. They attended the brief counseling session as a couple with the heavy drinker (their partner).
- Motivational Interviewing (MI) - Heavy Drinkers: People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. With their primary romantic partner, they attended three motivational interviewing sessions over a 60-day period. The sessions focused on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
- Motivational Interviewing (MI) - Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the MI arm. They attended the motivational interviewing sessions with the heavy drinker (their partner).
- Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers: People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. With their primary romantic partner, they attended three motivational interviewing sessions over a 60-day period. The sessions focused on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
  In addition to the counseling sessions, they received SMS messages twice per day prompting them to use a mobile app and a breathalyzer to test their blood alcohol levels (BAC). They received real-time feedback after each test.
- Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the MI Plus arm. In addition to attending the motivational interviewing sessions as a couple with the heavy drinker (their partner), they received real-time feedback about the drinker's BAC after each taken test and were alerted if the drinker missed a scheduled test.
Period: Overall Study
Arm/Group | Enhanced Usual Care- Heavy Drinkers | Enhanced Usual Care (EUC)- Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
Started | 31 | 31 | 31 | 31 | 31 | 31
Completed | 30 | 30 | 29 | 29 | 29 | 29
Not Completed | 1 | 1 | 2 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Ineligible | 0 | 0 | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Usual Care (EUC)- Heavy Drinkers: People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. They received the standard of care for alcohol use in addition to a brief alcohol counseling session modeled after WHO guidelines and Dr. Conroy's intervention in Malawi, which uses participants' baseline AUDIT scores for messaging around alcohol reduction and lasts 5-10 minutes. They attended this brief counseling session with their primary romantic partner.
  There were 31 people who were living with HIV and screened positive for heavy drinking assigned to this condition.
- Enhanced Usual Care (EUC) Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the EUC arm. They attended the brief counseling session as a couple with the heavy drinker (their partner).
- Motivational Interviewing (MI) - Heavy Drinkers: People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. With their primary romantic partner, they were to attend three motivational interviewing sessions over a 60-day period. The sessions focused on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
- Motivational Interviewing (MI) - Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the MI arm. In addition to attending the motivational interviewing sessions as a couple with the heavy drinker (their partner), they received real-time feedback about the drinker's BAC after each taken test and were alerted if the drinker missed a scheduled test.
  This group represents the romantic partners of the Heavy Drinkers assigned to the MI arm. 28 of these 30 participants also drank heavily. 15 were also living with HIV.
- Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners- Partner: These participants were the primary romantic partners of the heavy drinkers assigned to the MI Plus arm. In addition to attending the motivational interviewing sessions with the heavy drinker (their partner), they recieved real-time feedback about the drinker's BAC after each taken test and were alerted if the drinker missed a scheduled test.
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners- Partner | Total
Number analyzed (Participants) | 31 | 31 | 30 | 30 | 29 | 29 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.65 (6.69) | 38.39 (6.83) | 37.47 (7.51) | 35.73 (5.59) | 39.07 (6.42) | 36.62 (6.82) | 37.66 (6.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 23 | 14 | 16 | 8 | 21 | 90
  Male | 23 | 8 | 16 | 14 | 21 | 8 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 31 | 31 | 30 | 29 | 29 | 28 | 178
  White | 0 | 0 | 0 | 0 | 0 | 1 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 31 | 31 | 30 | 30 | 29 | 29 | 180
Score on Alcohol Use Disorders Identification Test (AUDIT) [Mean (Standard Deviation); unit: units on a scale (0-28).] — The AUDIT is a 10-item scale that assesses alcohol use and its consequences. The score is created by summing the responses to each of the items. Scores can range from 0-28. Higher scores indicate heavier/ riskier alcohol use.
  units on a scale (0-28). | 14.13 (6.02) | 9.84 (6.67) | 14.63 (6.60) | 11.57 (6.04) | 15.38 (6.18) | 14.03 (6.90) | 13.2 (6.6)
Number of participants who screened positive for heavy alcohol use [Count of Participants; unit: Participants] — At screening, we used the Alcohol Use Disorders Indentification Test- Consumption (AUDIT-C) to determine if a person was a heavy drinker. This is a three-item scale and scores range from 0 to 12. For men, a score of 4 or more indicates a likelihood of hazardous drinking. For women, the score to indicate a likelihood of hazardous drinking is 3 or more. Higher scores indicate riskier alcohol consumption.
  Participants | 31 | 26 | 30 | 28 | 29 | 26 | 170

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: Number of eligible individuals who enroll in the study
Time Frame: Baseline (Time 0)
Population: All couples who were eligible after screening enrolled in the study (i.e., engaged in the informed consent process, completed the baseline questionnaire, and were randomized). No one refused participation after randomization either.
Measure: Count of Participants; unit: Participants
Groups:
- Enhanced Usual Care (EUC)- Heavy Drinkers: People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. They received the standard of care for alcohol use in addition to a brief alcohol counseling session modeled after WHO guidelines and Dr. Conroy's intervention in Malawi, which uses participants' baseline AUDIT scores for messaging around alcohol reduction and lasts 5-10 minutes. They attended this brief counseling session with their primary romantic partner.
- Enhanced Usual Care (EUC) - Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the EUC arm. They attended the brief counseling session as a couple with the heavy drinker (their partner).
- Motivational Interviewing (MI)- Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the MI arm. They attended the motivational interviewing sessions with the heavy drinker (their partner).
- Motivatinal Interviewing Plus (MI Plus)- Heavy Drinkers: IPeople in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. With their primary romantic partner, they attended three motivational interviewing sessions over a 60-day period. The sessions focused on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
  In addition to the counseling sessions, they received SMS messages twice per day prompting them to use a mobile app and a breathalyzer to test their blood alcohol levels (BAC). They received real-time feedback after each test.
- Motivational Interviewing Plus (MI Plus)- Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the MI Plus arm. In addition to attending the motivational interviewing sessions with the heavy drinker (their partner), they received real-time feedback about the drinker's BAC after each taken test and were alerted if the drinker missed a scheduled test.
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI)- Partners | Motivatinal Interviewing Plus (MI Plus)- Heavy Drinkers | Motivational Interviewing Plus (MI Plus)- Partners
Number analyzed (Participants) | 31 | 31 | 30 | 30 | 29 | 29
Participants | 31 | 31 | 30 | 30 | 29 | 29

2. Primary Outcome: Retention Rate
Description: Number of enrolled individuals who completed the final follow-up survey (6-months post baseline)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Motivational Interviewing - Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the MI arm. They attended the motivational interviewing sessions with the heavy drinker (their partner).
- Motivational Interviewing Plus Breathalyzer (MI Plus)- Heavy Drinkers: People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. With their primary romantic partner, they attended three motivational interviewing sessions over a 60-day period. The sessions focused on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
  In addition to the counseling sessions, they received SMS messages twice per day prompting them to use a mobile app and a breathalyzer to test their blood alcohol levels (BAC). They received real-time feedback after each test.
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus)- Heavy Drinkers | Motivational Interviewing Plus (MI Plus)- Partners
Number analyzed (Participants) | 31 | 31 | 30 | 30 | 29 | 29
Participants | 30 | 30 | 29 | 29 | 29 | 29

3. Secondary Outcome: Satisfaction With Intervention
Description: number of participants who report being "satisfied" or "very satisfied" with the intervention at the two-month follow-up
Time Frame: 2 months
Population: We did not ask the participants in the Enhanced Usual Care arm about their satisfaction with the intervention. Two participants in the MI Heavy Drinkers and 2 participants in the MI Partners group did not complete the Time 2 survey, so were not asked these questions and not included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers: People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. With their primary romantic partner, they attended three motivational interviewing sessions over a 60-day period. The sessions focused on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
  In addition to the counseling sessions, they received SMS messages twice per day prompting them to use a mobile app and a breathalyzer to test their blood alcohol levels (BAC). They received real-time feedback after each test.
  Couples are made up of one person who is living with HIV and was identified during screening as a heavy drinker and his or her partner. The partner may or may be living with HIV and may or may not be a heavy drinker. The data presented includes both drinkers and thier partners. There were 29 couples (58 individuals) assigned to this arm.
- Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners: These participants were the primary romantic partners of the heavy drinkers assigned to the MI Plus arm. In addition to attending the motivational interviewing sessions with the heavy drinker (their partner), they received real-time feedback about the drinker's BAC after each taken test and were alerted if the drinker missed a scheduled test.
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
Number analyzed (Participants) | 0 | 0 | 28 | 28 | 29 | 29
Participants | 0 | 0 | 28 | 28 | 28 | 27

4. Secondary Outcome: Mid-point Survey Completion
Description: number of participants who complete the two-month survey
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- Motivational Interviewing (MI) - Heavy Drinkers: CPeople in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. With their primary romantic partner, they were to attend three motivational interviewing sessions over a 60-day period. The sessions focused on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
Number analyzed (Participants) | 31 | 31 | 30 | 30 | 29 | 29
Participants | 30 | 30 | 28 | 28 | 29 | 29

5. Secondary Outcome: Final Survey Completion
Description: number of couples who complete the six-month survey
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Motivational Interviewing Plus Breathalyzer (MI Plus): People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. With their primary romantic partner, they attended three motivational interviewing sessions over a 60-day period. The sessions focused on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
  In addition to the counseling sessions, they received SMS messages twice per day prompting them to use a mobile app and a breathalyzer to test their blood alcohol levels (BAC). They received real-time feedback after each test.
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
Number analyzed (Participants) | 31 | 31 | 30 | 30 | 29 | 29
Participants | 30 | 30 | 29 | 29 | 29 | 29

6. Secondary Outcome: Number of Participants Who Attended All Intervention Sessions
Description: Number of participants who attend all three intervention sessions
Time Frame: 2 months
Population: Participants in the Enhanced Usual Care Arm did were not assigned to any intervention sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
Number analyzed (Participants) | 0 | 0 | 30 | 30 | 29 | 29
Participants | 0 | 0 | 25 | 25 | 26 | 26

7. Secondary Outcome: 70% Breathalyzer Completion
Description: number of participants in the MI Plus - Heavy Drinker arm who complete 70% of breathalyzer tests
Time Frame: 2 months
Population: Only participants in the MI Plus- Heavy Drinker arm were given the breathalyzers and prompted to take tests
Measure: Count of Participants; unit: Participants
Groups:
- Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinker: People in this condition were living with HIV and screened positive for heavy drinking prior to enrollment. With their primary romantic partner, they attended three motivational interviewing sessions over a 60-day period. The sessions focused on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
  In addition to the counseling sessions, they received SMS messages twice per day prompting them to use a mobile app and a breathalyzer to test their blood alcohol levels (BAC). They received real-time feedback after each test.
Arm/Group | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinker
Number analyzed (Participants) | 29
Participants | 8

8. Secondary Outcome: Exploratory: ART Adherence
Description: Percentage of pills taken by HIV-infected participants in the past 30 days, using the bean count method (self-report) adapted from VAS
Time Frame: 6 months
Population: This analysis includes participants who were living with HIV and completed the 6-month follow-up survey.
Measure: Mean (Standard Deviation); unit: Percentage of pills taken
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
Number analyzed (Participants) | 29 | 22 | 29 | 15 | 29 | 19
Percentage of pills taken | 0.61 (0.44) | .91 (.19) | 0.70 (0.42) | .92 (.23) | 0.58 (0.45) | .89 (.23)

9. Secondary Outcome: Exploratory: Alcohol Use- Number of Drinking Days
Description: Number of drinking days in the past 30 days (self-report)
Time Frame: 6 months
Population: This analysis excluded participants who did not complete the 6-month follow-up survey. Data is missing for one participant in the EUC- partner condition.
Measure: Mean (Standard Deviation); unit: days out of the last 30
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
Number analyzed (Participants) | 30 | 29 | 29 | 29 | 29 | 29
days out of the last 30 | 8.2 (6.4) | 5.7 (6.3) | 6.3 (5.1) | 5.8 (5.6) | 7.9 (5.5) | 8.0 (6.5)

10. Secondary Outcome: Exploratory: Alcohol Use- Score on AUDIT at 2 Months
Description: Mean score on the Alcohol Use Disorders Identification Test- AUDIT prior 3 months. The AUDIT is a 10-item scale that assesses drinking behavior with a range of 0-40 (higher scores indicate higher alcohol use). A score of 8 or more may indicate hazardous or harmful drinking in both men and women.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
Number analyzed (Participants) | 30 | 30 | 28 | 28 | 29 | 29
units on a scale | 12.0 (6.2) | 10.43 (7.24) | 10.14 (5.94) | 11.11 (5.62) | 13.00 (6.82) | 11.38 (6.62)

11. Secondary Outcome: Exploratory: HIV Viral Load
Description: Number of HIV-infected index patients who are virally suppressed by local lab normal ranges, as measured by dried blood spots (DBS)
Time Frame: 2 months
Population: Viral load was only tested among heavy drinkers who completed the Time 2 follow-up
Measure: Count of Participants; unit: Participants
Groups:
- Enhanced Usual Care: Couples in this condition will receive the standard of care for alcohol use in addition to a brief alcohol counseling session modeled after WHO guidelines and Dr. Conroy's intervention in Malawi, which uses participants' baseline AUDIT scores for messaging around alcohol reduction and lasts 5-10 minutes.
  Couples are made up of one person who is living with HIV and was identified during screening as a heavy drinker and his or her partner. The partner may or may be living with HIV and may or may not be a heavy drinker. The data presented includes both drinkers and thier partners. There were 31 couples (62 individuals) assigned to this arm.
- Motivational Interviewing (MI): Couples will have three MI sessions over a 60-day period. These sessions will focus on communication between the couple, alcohol consumption patterns, and setting goals for alcohol-use reduction.
  Motivational Interviewing: Counseling
  Couples are made up of one person who is living with HIV and was identified during screening as a heavy drinker and his or her partner. The partner may or may be living with HIV and may or may not be a heavy drinker. The data presented includes both drinkers and thier partners. There were 30 couples (60 individuals) assigned to this arm.
- Motivational Interviewing Plus Breathalyzer (MI Plus): In addition to three MI sessions, drinkers in this condition will be prompted via SMS message twice per day to use a mobile app and a breathalyzer to test their blood alcohol levels (BAC). Both the drinker and their partner will receive real-time feedback about alcohol use.
  Motivational Interviewing: Counseling
  Motivational Interviewing plus Breathalyzer: Counseling plus mobile breathalyzer/ app
  Couples are made up of one person who is living with HIV and was identified during screening as a heavy drinker and his or her partner. The partner may or may be living with HIV and may or may not be a heavy drinker. The data presented includes both drinkers and thier partners. There were 29 couples (58 individuals) assigned to this arm.
Arm/Group | Enhanced Usual Care | Motivational Interviewing (MI) | Motivational Interviewing Plus Breathalyzer (MI Plus)
Number analyzed (Participants) | 30 | 29 | 29
Participants | 26 | 28 | 25

12. Secondary Outcome: Exploratory: Alcohol Use- Score on AUDIT at 6 Months
Description: as for outcome 10
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
Number analyzed (Participants) | 30 | 30 | 29 | 29 | 29 | 29
units on a scale | 7.83 (4.83) | 9.93 (6.41) | 8.80 (6.77) | 10.62 (5.82) | 8.27 (5.81) | 11.07 (7.21)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year.
Description: Our definition did not vary from clinicaltrials.gov. We collected information about adverse events during data collection and during calls to participants regarding scheduled visits.
Arm/Group | Enhanced Usual Care (EUC)- Heavy Drinkers | Enhanced Usual Care (EUC) - Partners | Motivational Interviewing (MI) - Heavy Drinkers | Motivational Interviewing (MI) - Partners | Motivational Interviewing Plus Breathalyzer (MI Plus) - Heavy Drinkers | Motivational Interviewing Plus Breathalyzer (MI Plus) - Partners
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/30 | 0/30 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/30 | 0/30 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/30 | 0/30 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT05756790/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT05756790/ICF_001.pdf